CLINICAL TRIAL: NCT01312779
Title: Clinical Evaluation of the Size 23mm Carpentier-Edwards PERIMOUNT Magna Mitral Bioprosthesis, Model 7000TFX
Brief Title: Magna Mitral - 23mm
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Edwards Lifesciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2008-07
Record Dates: First submitted 2011-03-09; First posted 2011-03-11 (Estimated); Results first posted 2020-03-03 (Actual); Last update posted 2020-03-18 (Actual); Status verified 2020-03

CONDITIONS: Mitral Heart Valve Disease
Keywords: Mitral Valve Replacement; 23mm CEP; Magna
MeSH Terms: conditions — Heart Valve Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- All subjects receive implant (Other): Subjects serve as own control
  Interventions: Device: Implantation of CEP Magna Mitral Model 7000TFX

INTERVENTIONS:
Device: Implantation of CEP Magna Mitral Model 7000TFX — Heart valve surgery: CEP Magna Mitral Model 7000 TFX

SUMMARY:
The purpose of this clinical study is to obtain human clinical data that demonstrates that the size 23mm Carpentier-Edwards PERIMOUNT Magna mitral pericardial valve, model 7000TFX, is a safe and effective replacement heart valve.

DETAILED DESCRIPTION:
This is a prospective, non-randomized, multi-site, descriptive study. A minimum of 15 and up to 20 subjects will be implanted at a minimum of 2 and up to 8 participating investigational sites within the US and internationally.

ELIGIBILITY:
Inclusion Criteria:

1. Patient has mitral valve disease requiring surgical replacement
2. Patient has provided written informed consent prior to mitral valve surgery
3. Patient is expected to survive surgery and be discharged
4. Patient is willing to comply with specified follow-up evaluations
5. Patient is 13 years of age or older

Exclusion Criteria:

1. Patient has life expectancy < 12 months due to non-cardiac co-morbid conditions;
2. Patient has/had active endocarditis within the last 3 months
3. Patient requires replacement of a native or previously implanted prosthetic, tricuspid, pulmonic or aortic valve;
4. Patient was previously enrolled and implanted in the study
5. Patient has/had prior aortic, tricuspid and/ or pulmonary valve surgery, which included implantation of a bioprosthetic valve or mechanical valve that will remain in situ
6. Patient has a body surface area (BSA) > 1.9m2
7. Female patients who are pregnant, planning to become pregnant, or lactating
8. Patient has a documented history of substance ( drug or alcohol) abuse
9. Patient is currently a prison inmate
10. Patient is currently participating in an investigational drug or another device study
11. Patient is undergoing renal dialysis for chronic renal failure or has hyperparathyroidism
12. Patient has active myocarditis
13. Patient has had an acute preoperative neurological deficit, myocardial infarction, or cardiac event and has not returned to baseline or stabilized > 30 days prior to the planned v alve implant surgery
14. Patient has an abnormality such as an aortic aneurysm (e.g. due to cystic medial necrosis or Marfan's syndrome), aortic dissection, or ventricular aneurysm that might place

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2011-03 (Actual); Primary Completion 2018-11 (Actual); Study Completion 2018-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (6):
- United States (5):
  - Florida Hospital, Orlando, Florida
  - Northwestern Hospital, Chicago, Illinois
  - University of Iowa Hospitals & Clinics, Iowa City, Iowa
  - Washington University, St Louis, Missouri
  - Cooper University Hospital, Camden, New Jersey
- The John Paul II Hospital in Krakow, Krakow, Poland

REFERENCES:
- See also: New York Heart Association Classification — https://www.heart.org/en/health-topics/heart-failure/what-is-heart-failure/classes-of-heart-failure

RESULTS

PARTICIPANT FLOW:
Groups:
- Magna Mitral 23: Clinical Evaluation of the size 23 mm Carpentier-Edwards PERIMOUNT Magna Mitral Bioprosthesis, Model 7000TFX
Period: Overall Study
Arm/Group | Magna Mitral 23
Started | 39
Implanted With Device | 12
Completed | 7
Not Completed | 32
Not completed — Withdrawal by Subject | 2
Not completed — Death | 3
Not completed — Not Implanted with Device | 27

BASELINE CHARACTERISTICS:
Population: The outcome is reported for subjects who received the Magna Mitral, Model 7000TFX device where data is available.
Arm/Group | Magna Mitral 23
Number analyzed (Participants) | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.5 (14.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Percent of Early Adverse Events Divided
Description: Number of early adverse events occurring within 30 days of procedure divided by the number of enrolled subjects times 100.
Time Frame: Events occuring within 30 days of procedure
Population: The outcome is reported for subjects who received the Magna Mitral, Model 7000TFX device where data is available.
Measure: Number; unit: percentage of subjects
Arm/Group | Magna Mitral 23
Number analyzed (Participants) | 12
percentage of subjects
  Death | 8.3
  Valve-Related Death | 0.0
  Thromboembolism | 0.0
  Valve Thrombosis | 0.0
  Hemorrhage | 0.0
  Major Hemorrhage | 0.0
  Non-Structural Valve Dysfunction (study valve) | 8.3
  All Clinically Significant PVL | 8.3
  Major Clinically Significant PVL | 0.0
  Hemolysis | 0.0
  Endocarditis | 0.0
  Structural Valve Deterioration | 0.0
  Reoperation | 0.0
  Explant | 0.0

2. Primary Outcome: Percent of Late Adverse Events
Description: Number of late events divided by the total number of late patient years times 100. Late patient years are calculated from 31 days post-implant to the date of the last contact (follow up or adverse event).
Time Frame: Events occurring >= 31 days and up through 5 years post-implant
Population: The outcome is reported for subjects who received the Magna Mitral, Model 7000TFX device where data is available.
Measure: Number; unit: percentage of events/late patient years
Arm/Group | Magna Mitral 23
Number analyzed (Participants) | 11
percentage of events/late patient years
  Death | 4.5
  Valve-Related Death | 2.2
  Thromboembolism | 2.2
  Valve Thrombosis | 0.0
  Hemorrhage | 2.2
  Major Hemorrhage | 2.2
  Non-Structural Valve Dysfunction (study valve) | 0.0
  All Clinically Significant PVL | 0.0
  Major Clinically Significant PVL | 0.0
  Hemolysis | 0.0
  Endocarditis | 2.2
  Structural Valve Deterioration | 6.7
  Reoperation | 6.7
  Explant | 6.7

3. Primary Outcome: Percentage of Subjects With Freedom From Serious Adverse Events (SAE) Post-implant > 30 Days
Description: Subject's freedom from Serious Adverse Events at > 30 days post-implant. Time to events were estimated by Kaplan-Meier method.
Time Frame: >30 Days, 1 Year, 2 Years, 3 Years, 4 Years, and 5 Years post-implant
Population: The outcome is reported for subjects who received the Magna Mitral, Model 7000TFX device where data is available.
Measure: Number; unit: percentage of subjects
Groups:
- Magna Mitral 23 - >30 Days Post-implant; Magna Mitral 23 - 1 Year Post-implant; Magna Mitral 23 - 2 Years Post-implant; Magna Mitral 23 - 3 Years Post-implant; Magna Mitral 23 - 4 Years Post-implant; Magna Mitral 23 - 5 Years Post-implant: Clinical Evaluation of the size 23 mm Carpentier-Edwards PERIMOUNT Magna Mitral Bioprosthesis, Model 7000TFX
Arm/Group | Magna Mitral 23 - >30 Days Post-implant | Magna Mitral 23 - 1 Year Post-implant | Magna Mitral 23 - 2 Years Post-implant | Magna Mitral 23 - 3 Years Post-implant | Magna Mitral 23 - 4 Years Post-implant | Magna Mitral 23 - 5 Years Post-implant
Number analyzed (Participants) | 11 | 11 | 11 | 11 | 11 | 11
percentage of subjects
  Death | 100.00 | 90.91 | 90.91 | 90.91 | 80.81 | 80.81
  Valve-related Death | 100.00 | 100.0 | 100.0 | 100.0 | 88.89 | 88.89
  Reoperation | 100.00 | 100.00 | 100.00 | 100.00 | 100.00 | 87.50
  Explant | 100.00 | 100.00 | 100.00 | 100.00 | 100.00 | 87.50
  Bleeding Event | 100.00 | 90.00 | 90.00 | 90.00 | 90.00 | 90.00
  Major Bleeding Event | 100.00 | 90.00 | 90.00 | 90.00 | 90.00 | 90.00
  Thromboembolism | 100.00 | 100.00 | 88.89 | 88.89 | 88.89 | 88.89
  Endocarditis | 100.00 | 100.00 | 100.00 | 100.00 | 88.89 | 88.89
  Perivalvular Leak | 100.00 | 100.00 | 100.00 | 100.00 | 100.00 | 100.00
  Major Perivalvular Leak | 100.00 | 100.00 | 100.00 | 100.00 | 100.00 | 100.00
  Hemolysis | 100.00 | 100.00 | 100.00 | 100.00 | 100.00 | 100.00
  Non-structural Valve Dysfunction | 100.00 | 100.00 | 100.00 | 100.00 | 100.00 | 100.00
  Structural Valve Deterioration | 100.00 | 100.00 | 100.00 | 100.00 | 100.00 | 87.50
  Valve Thrombosis | 100.00 | 100.00 | 100.00 | 100.00 | 100.00 | 100.00

4. Primary Outcome: Subject's Average Effective Orifice Area (EOA) Measurement
Description: Effective orifice area represents the cross-sectional area of the blood flow downstream of the mitral valve. Effective orifice area is evaluated by echocardiography over time.
Time Frame: Pre-procedure and 1 Year post-Implant
Population: The outcome is reported for subjects who received the Magna Mitral, Model 7000TFX device where data is available.
Measure: Mean (Standard Deviation); unit: Centimeters Squared
Arm/Group | Magna Mitral 23
Number analyzed (Participants) | 12
Centimeters Squared
  Pre-Procedure: number analyzed (Participants) | 4
  Pre-Procedure | 0.8 (0.2)
  1 Year: number analyzed (Participants) | 8
  1 Year | 1.2 (0.2)

5. Other Pre Specified Outcome: Subject's Average Mean Gradient Measurement
Description: Mean gradient is the average flow of blood through the mitral valve measured in millimeters of mercury. Gradients are evaluated by echocardiography over time. Mean gradient values depend on the size and type of valve.
Time Frame: Pre-procedure and 1 Year post-implant
Population: The outcome is reported for subjects who received the Magna Mitral, Model 7000TFX device where data is available.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Magna Mitral 23
Number analyzed (Participants) | 12
mmHg
  Pre-Procedure: number analyzed (Participants) | 10
  Pre-Procedure | 9.8 (5.3)
  1 Year: number analyzed (Participants) | 9
  1 Year | 7.5 (1.7)

6. Other Pre Specified Outcome: Subject's Average Peak Gradient Measurement
Description: Peak gradient is the maximum value measured of flow of blood through the mitral valve as measured in millimeters of mercury. Gradients are evaluated by echocardiography over time.
Time Frame: Pre-procedure and 1 Year post-implant
Population: The outcome is reported for subjects who received the Magna Mitral, Model 7000TFX device where data is available.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Magna Mitral 23
Number analyzed (Participants) | 12
mmHg
  Pre-Procedure: number analyzed (Participants) | 10
  Pre-Procedure | 19.1 (7.5)
  1 Year: number analyzed (Participants) | 9
  1 Year | 16.8 (5.1)

7. Other Pre Specified Outcome: Subject's Average Effective Orifice Area Index (EOAI) Measurement
Description: Effective orifice area index represents the minimal cross-sectional area of the blood flow downstream of the mitral valve divided by the person's body surface area. Effective orifice area index is evaluated by echocardiography over time.
Time Frame: Pre-procedure and 1 Year post-implant
Population: The outcome is reported for subjects who received the Magna Mitral, Model 7000TFX device where data is available.
Measure: Mean (Standard Deviation); unit: cm^2/m^2
Arm/Group | Magna Mitral 23
Number analyzed (Participants) | 12
cm^2/m^2
  Pre-Procedure: number analyzed (Participants) | 4
  Pre-Procedure | 0.5 (0.1)
  1 Year: number analyzed (Participants) | 8
  1 Year | 0.7 (0.1)

8. Other Pre Specified Outcome: Subject's Average Performance Index Measurement
Description: Performance index is defined as the subject's effective orifice area (the cross sectional area of the blood flow downstream of the mitral valve) divided by the subject's native orifice area. Effective orifice area is evaluated by echocardiography over time.
Time Frame: Pre-procedure and 1 Year post-Implant
Population: The outcome is reported for subjects who received the Magna Mitral, Model 7000TFX device where data is available.
Measure: Mean (Standard Deviation); unit: cm^2/cm^2
Arm/Group | Magna Mitral 23
Number analyzed (Participants) | 12
cm^2/cm^2
  Pre-Procedure: number analyzed (Participants) | 4
  Pre-Procedure | 0.7 (0.2)
  1 Year: number analyzed (Participants) | 8
  1 Year | 1.0 (0.1)

9. Other Pre Specified Outcome: Subject's Average Cardiac Output
Description: The amount of blood the heart pumps through the circulatory system in a minute.
Time Frame: Pre-procedure and 1 Year post-implant
Population: The outcome is reported for subjects who received the Magna Mitral, Model 7000TFX device where data is available.
Measure: Mean (Standard Deviation); unit: Liters/minute
Arm/Group | Magna Mitral 23
Number analyzed (Participants) | 12
Liters/minute
  Pre-Procedure: number analyzed (Participants) | 10
  Pre-Procedure | 4.0 (0.8)
  1 Year: number analyzed (Participants) | 9
  1 Year | 4.8 (0.7)

10. Other Pre Specified Outcome: Subject's Average Cardiac Index
Description: Cardiac index is an assessment that divides the cardiac output from the left ventricle in one minute by the person's body surface area (BSA), thus relating heart performance to the size of the individual.
Time Frame: Pre-procedure and 1 Year post-implant
Population: The outcome is reported for subjects who received the Magna Mitral, Model 7000TFX device where data is available.
Measure: Mean (Standard Deviation); unit: L/min/m2
Arm/Group | Magna Mitral 23
Number analyzed (Participants) | 12
L/min/m2
  Pre-Procedure: number analyzed (Participants) | 10
  Pre-Procedure | 2.4 (0.4)
  1 Year: number analyzed (Participants) | 9
  1 Year | 2.9 (0.5)

11. Other Pre Specified Outcome: Subject's Average Left Ventricular Mass Regression
Description: Patients can experience an enlargement of the left ventricle (chamber) of their heart because it works harder with a defective heart valve. Left ventricular mass regression evaluates if the patient experiences a decrease in the size of the left ventricle (chamber) after the repair or replacement of their heart valve.
Time Frame: Pre-procedure and 1 Year post-implant
Population: The outcome is reported for subjects who received the Magna Mitral, Model 7000TFX device where data is available.
Measure: Mean (Standard Deviation); unit: grams
Arm/Group | Magna Mitral 23
Number analyzed (Participants) | 12
grams
  Pre-Procedure: number analyzed (Participants) | 10
  Pre-Procedure | 161.0 (42.4)
  1 Year: number analyzed (Participants) | 9
  1 Year | 130.7 (35.1)

12. Other Pre Specified Outcome: Subject's Severity of Central Mitral Regurgitation at 1 Year Post-implant.
Description: Mitral valvular regurgitation occurs when the mitral valve in the heart does not close tightly allowing some of the blood that was pumped out of the heart to leak back into it. Mitral valvular regurgitation is evaluated by echocardiography over time. It is assessed on a scale from 0 to 4, where 0 represents no regurgitation and 4 represents severe regurgitation.
Time Frame: 1 Year post-implant
Population: The outcome is reported for subjects who received the Magna Mitral, Model 7000TFX device where data is available.
Measure: Count of Participants; unit: Participants
Arm/Group | Magna Mitral 23
Number analyzed (Participants) | 9
Participants
  None | 3
  +1 Trivial/Trace | 5
  +2 Mild | 1
  +3 Modearte | 0
  +4 Severe | 0

13. Other Pre Specified Outcome: Subject's Average Red Blood Cells Count
Description: Laboratory Analysis of Red Blood Cell (RBC) Count on blood drawn from subjects; RBC carry oxygen.
Time Frame: Baseline, 6 Month, 1 Year, 2 Years, 3 Years, 4 Years, and 5 Years post-implant
Population: The outcome is reported for subjects who received the Magna Mitral, Model 7000TFX device where data is available.
Measure: Mean (Standard Deviation); unit: 10^6 cells/microliters
Arm/Group | Magna Mitral 23
Number analyzed (Participants) | 12
10^6 cells/microliters
  Baseline | 4.1 (0.7)
  6 Month: number analyzed (Participants) | 8
  6 Month | 4.4 (0.9)
  1 Year: number analyzed (Participants) | 9
  1 Year | 4.4 (0.3)
  2 Year: number analyzed (Participants) | 9
  2 Year | 4.1 (0.6)
  3 Year: number analyzed (Participants) | 9
  3 Year | 3.9 (1.0)
  4 Year: number analyzed (Participants) | 8
  4 Year | 4.1 (0.6)
  5 Year: number analyzed (Participants) | 7
  5 Year | 4.0 (0.6)

14. Other Pre Specified Outcome: Subject's Average White Blood Cell Count
Description: Laboratory analysis of White Blood Cell (WBC) Count on blood drawn from subject; WBC fight infection.
Time Frame: Baseline, 6 Month, 1 Year, 2 Years, 3 Years, 4 Years, and 5 Years post-implant
Population: The outcome is reported for subjects who received the Magna Mitral, Model 7000TFX device where data is available.
Measure: Mean (Standard Deviation); unit: 10^3 cells /microliter
Arm/Group | Magna Mitral 23
Number analyzed (Participants) | 12
10^3 cells /microliter
  Baseline | 7.1 (1.7)
  6 Month: number analyzed (Participants) | 8
  6 Month | 7.5 (2.4)
  1 Year: number analyzed (Participants) | 9
  1 Year | 7.4 (2.3)
  2 Year: number analyzed (Participants) | 9
  2 Year | 7.4 (1.8)
  3 Year: number analyzed (Participants) | 9
  3 Year | 7.1 (1.8)
  4 Year: number analyzed (Participants) | 8
  4 Year | 8.9 (3.0)
  5 Year: number analyzed (Participants) | 7
  5 Year | 7.1 (1.4)

15. Other Pre Specified Outcome: Subject's Average Hematocrit Percentage
Description: Laboratory Analysis of Hematocrit Percentage on blood drawn from subjects. Hematocrit is the proportion of red blood cells to the plasma (liquid portion of the blood).
Time Frame: Baseline, 6 Month, 1 Year, 2 Years, 3 Years, 4 Years, and 5 Years post-implant
Population: The outcome is reported for subjects who received the Magna Mitral, Model 7000TFX device where data is available.
Measure: Mean (Standard Deviation); unit: percentage of red blood cells
Arm/Group | Magna Mitral 23
Number analyzed (Participants) | 12
percentage of red blood cells
  Baseline | 38.3 (6.0)
  6 Month: number analyzed (Participants) | 8
  6 Month | 40.6 (6.6)
  1 Year: number analyzed (Participants) | 9
  1 Year | 41.2 (3.4)
  2 Year: number analyzed (Participants) | 9
  2 Year | 39.7 (4.3)
  3 Year: number analyzed (Participants) | 9
  3 Year | 36.3 (7.0)
  4 Year: number analyzed (Participants) | 8
  4 Year | 40.1 (4.0)
  5 Year: number analyzed (Participants) | 7
  5 Year | 37.4 (3.7)

16. Other Pre Specified Outcome: Subject's Average Plasma Free Hemoglobin
Description: Laboratory Analysis of Plasma Free Hemoglobin on blood drawn from subjects. This blood test measures the level of free hemoglobin in the plasma (liquid portion of the blood).
Time Frame: Baseline, 6 Month, 1 Year, 2 Years, 3 Years, 4 Years, and 5 Years post-implant
Population: The outcome is reported for subjects who received the Magna Mitral, Model 7000TFX device where data is available.
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Magna Mitral 23
Number analyzed (Participants) | 12
mg/dl
  Baseline: number analyzed (Participants) | 9
  Baseline | 12.9 (13.9)
  6 Month: number analyzed (Participants) | 5
  6 Month | 23.1 (19.5)
  1 Year: number analyzed (Participants) | 8
  1 Year | 11.2 (11.8)
  2 Year: number analyzed (Participants) | 6
  2 Year | 14.8 (9.2)
  3 Year: number analyzed (Participants) | 4
  3 Year | 5.1 (3.4)
  4 Year: number analyzed (Participants) | 4
  4 Year | 22.3 (15.6)
  5 Year: number analyzed (Participants) | 3
  5 Year | 9.9 (9.4)

17. Other Pre Specified Outcome: Subject's Average Hemoglobin Count
Description: Laboratory Analysis of Hemoglobin Count on blood drawn from subjects. Hemoglobin is an oxygen-carrying protein in red blood cells.
Time Frame: Baseline, 6 Month, 1 Year, 2 Years, 3 Years, 4 Years, and 5 Years post-implant
Population: The outcome is reported for subjects who received the Magna Mitral, Model 7000TFX device where data is available.
Measure: Mean (Standard Deviation); unit: g/dl
Arm/Group | Magna Mitral 23
Number analyzed (Participants) | 12
g/dl
  Baseline | 12.5 (2.1)
  6 Month: number analyzed (Participants) | 8
  6 Month | 13.3 (2.3)
  1 Year: number analyzed (Participants) | 9
  1 Year | 13.5 (1.5)
  2 Year: number analyzed (Participants) | 9
  2 Year | 13.0 (1.7)
  3 Year: number analyzed (Participants) | 9
  3 Year | 12.1 (2.6)
  4 Year: number analyzed (Participants) | 8
  4 Year | 13.4 (1.7)
  5 Year: number analyzed (Participants) | 7
  5 Year | 12.1 (1.5)

18. Other Pre Specified Outcome: Subject's Average Platelet Count
Description: Laboratory Analysis of Platelet Count on blood drawn from subjects; platelets help with blood clotting.
Time Frame: Baseline, 6 Month, 1 Year, 2 Years, 3 Years, 4 Years, and 5 Years post-implant
Population: The outcome is reported for subjects who received the Magna Mitral, Model 7000TFX device where data is available.
Measure: Mean (Standard Deviation); unit: 10^3 platelets per microliter
Arm/Group | Magna Mitral 23
Number analyzed (Participants) | 12
10^3 platelets per microliter
  Baseline | 244.8 (95.6)
  6 Months: number analyzed (Participants) | 8
  6 Months | 231.1 (77.7)
  1 Year: number analyzed (Participants) | 9
  1 Year | 199.7 (39.5)
  2 Year: number analyzed (Participants) | 9
  2 Year | 201.8 (63.8)
  3 Year: number analyzed (Participants) | 9
  3 Year | 217.9 (78.0)
  4 Year: number analyzed (Participants) | 8
  4 Year | 236.3 (98.8)
  5 Year: number analyzed (Participants) | 7
  5 Year | 208.6 (71.8)

19. Other Pre Specified Outcome: Number and Percentage of Subjects in NYHA Functional Class I or II at 1 Year Post-Implant.
Description: The New York Heart Association (NYHA) functional classification system relates symptoms to everyday activities and the patient's quality of life.
  Class I. No limitation of physical activity. Ordinary physical activity does not cause undue fatigue, palpitation, dyspnea (shortness of breath).
  Class II. Slight limitation of physical activity. Comfortable at rest. Ordinary physical activity results in fatigue, palpitation, dyspnea (shortness of breath).
Time Frame: Baseline and 1 Year post-implant
Population: The outcome is reported for subjects who received the Magna Mitral, Model 7000TFX device where data is available.
Measure: Count of Participants; unit: Participants
Groups:
- Baseline NYHA - Magna Mitral 23; 1 Year NYHA - Magna Mitral 23: Clinical Evaluation of the size 23 mm Carpentier-Edwards PERIMOUNT Magna Mitral Bioprosthesis, Model 7000TFX
Arm/Group | Baseline NYHA - Magna Mitral 23 | 1 Year NYHA - Magna Mitral 23
Number analyzed (Participants) | 12 | 9
Participants
  Class I | 1 | 7
  Class II | 5 | 1

20. Other Pre Specified Outcome: Subject's New York Heart Association (NYHA) Functional Class Compared to Baseline
Description: The New York Heart Association (NYHA) functional classification system relates symptoms to everyday activities and the patient's quality of life.
  Class I. No limitation of physical activity. Ordinary physical activity does not cause undue fatigue, palpitation, dyspnea (shortness of breath).
  Class II. Slight limitation of physical activity. Comfortable at rest. Ordinary physical activity results in fatigue, palpitation, dyspnea (shortness of breath).
  Class III. Marked limitation of physical activity. Comfortable at rest. Less than ordinary activity causes fatigue, palpitation, or dyspnea.
  Class IV. Unable to carry on any physical activity without discomfort. Symptoms of heart failure at rest. If any physical activity is undertaken, discomfort increases.
Time Frame: 6 Months, 1 Year, 2 Years, 3 Years, 4 Years, and 5 Years post-implant
Population: The outcome is reported for subjects who received the Magna Mitral, Model 7000TFX device where data is available.
Measure: Count of Participants; unit: Participants
Arm/Group | Magna Mitral 23
Number analyzed (Participants) | 12
Participants
  6 Months: number analyzed (Participants) | 9
  6 Months: Improved | 7
  6 Months: Same | 2
  6 Months: Worsened | 0
  1 Year: number analyzed (Participants) | 9
  1 Year: Improved | 8
  1 Year: Same | 1
  1 Year: Worsened | 0
  2 Year: number analyzed (Participants) | 9
  2 Year: Improved | 7
  2 Year: Same | 2
  2 Year: Worsened | 0
  3 Year: number analyzed (Participants) | 9
  3 Year: Improved | 7
  3 Year: Same | 1
  3 Year: Worsened | 1
  4 Year: number analyzed (Participants) | 8
  4 Year: Improved | 5
  4 Year: Same | 2
  4 Year: Worsened | 1
  5 Year: number analyzed (Participants) | 7
  5 Year: Improved | 3
  5 Year: Same | 2
  5 Year: Worsened | 2

21. Other Pre Specified Outcome: Subject's Average Score on the EQ-5D- Quality of Life Questionnaire Over Time
Description: The EQ-5D is a standardized questionnaire that asks subjects to rate themselves (no problems, some problems, extreme problems) on mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. The scale is indexed and ranges from a minimum of 0.275 and a maximum of 1.000. A lower number indicates the participants experiences more problems and a higher number indicates the participants experiences fewer problems.
Time Frame: 6 Months and 1 Year post-implant
Population: The outcome is reported for subjects who received the Magna Mitral, Model 7000TFX device where data is available.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- EQ-5D at Baseline: EQ-5D data.Clinical Evaluation of the size 23 mm Carpentier-Edwards PERIMOUNT Magna Mitral Bioprosthesis, Model 7000TFX
Arm/Group | EQ-5D at Baseline
Number analyzed (Participants) | 12
units on a scale
  Baseline: number analyzed (Participants) | 9
  Baseline | 0.86 (0.07)
  6 Month: number analyzed (Participants) | 9
  6 Month | 0.94 (0.07)
  1 Year: number analyzed (Participants) | 9
  1 Year | 0.89 (0.11)

ADVERSE EVENTS:
Time Frame: Events occurring from baseline through five years post implant
Description: The outcome is reported for subjects who received the Magna Mitral, Model 7000TFX device where data is available.
Arm/Group | Magna Mitral 23
All-Cause Mortality (participants affected / at risk) | 3/12
Serious Adverse Events (participants affected / at risk) | 12/12
Other Adverse Events (participants affected / at risk) | 11/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Magna Mitral 23 (N=12)
Heart Failure - Acute (Cardiac disorders) | 5 (6)
Gastrointestinal - Other (Gastrointestinal disorders) | 3 (5)
Heart Failure - Chronic (CHF) (Cardiac disorders) | 4 (4)
Cancer - Newly Diagnosed (General disorders) | 3 (4)
Miscellaneous Complication (General disorders) | 3 (4)
Neurologic - Other (Psychiatric disorders) | 3 (4)
Respiratory Infection - Pneumonia (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Other Infection/Inflammation (Respiratory, thoracic and mediastinal disorders) | 1 (3)
Arrhythmia - AV Block (Cardiac disorders) | 2 (2)
Respiratory Dysfunction/Insufficiency (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Anemia - Non-Bleeding Related (Blood and lymphatic system disorders) | 1 (1)
Angina, Unstable (Cardiac disorders) | 1 (1)
Arrhythmia - Atrial Flutter (Cardiac disorders) | 1 (1)
Arrhythmia - Paroxysmal Atrial Fibrillation (PAF) (Cardiac disorders) | 1 (1)
Biliary (Gallbladder) (Gastrointestinal disorders) | 1 (1)
Bleeding - Cardiovascular (Blood and lymphatic system disorders) | 1 (1)
Cardiogenic Shock (Cardiac disorders) | 1 (1)
Cardiovascular Other (Cardiac disorders) | 1 (1)
Endocarditis (Cardiac disorders) | 1 (1)
Endocrine Complications (Gastrointestinal disorders) | 1 (1)
Gastrointestinal - Infection (Diarrhea) (Gastrointestinal disorders) | 1 (1)
Neurologic - Dizziness (Psychiatric disorders) | 1 (1)
Non Structural Valve Dysfunction (NSVD) - Non-Perivalvular Leak (Cardiac disorders) | 1 (1)
Psychiatric Disorder (Psychiatric disorders) | 1 (1)
Pulmonary Edema (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary Hypertension (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Structural Valve Deterioration (SVD) (Cardiac disorders) | 1 (1)
Thromboembolic Event - Transient Ischemic Attack (TIA) (Cardiac disorders) | 1 (1)
Vascular - Other (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Magna Mitral 23 (N=12)
Miscellaneous Complication (General disorders) | 6 (12)
Thrombocytopenia - Non-Heparin Induced (Blood and lymphatic system disorders) | 5 (7)
Gastrointestinal - Other (Gastrointestinal disorders) | 5 (6)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 5 (6)
Respiratory Infection - Upper (URI) (Respiratory, thoracic and mediastinal disorders) | 5 (6)
Anemia - Bleeding Related (Blood and lymphatic system disorders) | 4 (6)
Skin/Skeletal/Other (Respiratory, thoracic and mediastinal disorders) | 4 (6)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 4 (5)
Anemia - Non-Bleeding Related (Blood and lymphatic system disorders) | 4 (4)
Arrhythmia - Atrial Fibrillation (Cardiac disorders) | 4 (4)
Arrhythmia - Bradycardia (Cardiac disorders) | 4 (4)
Urinary Tract Infection (UTI) (Renal and urinary disorders) | 4 (4)
Blood/Lymphatic/Other (Blood and lymphatic system disorders) | 3 (3)
Respiratory Dysfunction/Insufficiency (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Arrhythmia - Bundle Branch Block (Cardiac disorders) | 2 (3)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Other Infection/Inflammation (Respiratory, thoracic and mediastinal disorders) | 1 (3)
Arrhythmia - Atrial Flutter (Cardiac disorders) | 2 (2)
Cardiovascular Other (Cardiac disorders) | 2 (2)
Gastrointestinal - Infection (Diarrhea) (Gastrointestinal disorders) | 2 (2)
Heart Failure - Acute (Cardiac disorders) | 2 (2)
Hypotension (Cardiac disorders) | 2 (2)
Neurologic - Dizziness (Psychiatric disorders) | 2 (2)
Neurologic - Other (Psychiatric disorders) | 2 (2)
Renal - Other (Renal and urinary disorders) | 2 (2)
Arrhythmia - AV Block (Cardiac disorders) | 1 (1)
Arrhythmia - Tachy-Bradycardia (Cardiac disorders) | 1 (1)
Arrhythmia - Tachycardia (Cardiac disorders) | 1 (1)
Bleeding - Cardiovascular (Blood and lymphatic system disorders) | 1 (1)
Bleeding - Peripheral Vascular (E.G. Nosebleeds; Hematomas) (Blood and lymphatic system disorders) | 1 (1)
Cancer - Newly Diagnosed (General disorders) | 1 (1)
Cancer - Progression Of Underlying Disease (General disorders) | 1 (1)
Endocrine Complications (Gastrointestinal disorders) | 1 (1)
Hepatic - Complication (Gastrointestinal disorders) | 1 (1)
Minor (<=+2) Paravalvular Leak (Cardiac disorders) | 1 (1)
Neurologic - Syncope (Psychiatric disorders) | 1 (1)
Pulmonary/Respiratory Other (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory Infection - Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Thrombocytopenia - Heparin Induced (HIT) (Blood and lymphatic system disorders) | 1 (1)
Transient Psychotic Syndrome (Psychiatric disorders) | 1 (1)
Vaginal Infection (Renal and urinary disorders) | 1 (1)
Valve - Other (Cardiac disorders) | 1 (1)
Vascular - Other (Vascular disorders) | 1 (1)
Vision Disorder (General disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Publication of overall study results which have not been released requires written approval of Sponsor, but presentation of site-specific results can occur subject to review by Sponsor. Manuscripts will be submitted to Sponsor for review 30 days prior to submission of manuscript for publication/presentation. Sponsor may ask for a 60 day delay of submission of manuscripts for publication to protect proprietary information and filing of related patent applications.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2011-11-11): https://cdn.clinicaltrials.gov/large-docs/79/NCT01312779/Prot_SAP_000.pdf